CLINICAL TRIAL: NCT01222481
Title: A Comprehensive Assessment of Adult Head and Neck Cancer Survivors (A Pilot Study)
Brief Title: Comprehensive Assessment of Head and Neck Cancer Survivors
Acronym: CAHNCA
Status: Completed | Type: Observational
Sponsor: Jay F. Piccirillo, MD (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor-Investigator, Jay F. Piccirillo, MD, Professor, Washington University School of Medicine, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: 09-0433
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Functional Status; Cognitive Status; Neurocognitive Assessments; Performance-based Assessments; Cancer; Function; Cognition; Quality of Life
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newly-diagnosed Head and Neck Cancer

SUMMARY:
Cancer survivorship has dramatically improved within the last four decades and a greater number of Americans are living after cancer diagnosis. An increase in the number of survivors has highlighted the need to investigate the quality of life experienced by these survivors. While Survivorship research has improved our understanding of the challenges faced by some cancer survivors, there is a paucity of research on the functional and cognitive health status of head and neck cancer survivors.

The purpose of this study is to evaluate the functional and cognitive changes that occur in head and neck cancer patients as a result of cancer treatment, in an attempt to increase our understanding of the complex interactions between cancer treatment, comorbid health ailments and quality of life.

DETAILED DESCRIPTION:
Cancer is the second leading cause of death in the United States today, accounting for nearly a quarter of total deaths. Due to advancements in cancer management, specifically in the areas of surveillance, early diagnosis, and utilization of evidenced-based therapies, there has been an increase in the number of survivors in the United States. As at 2007, there were over 11 million cancer survivors in the United States and this number is projected to reach 15 million by the end of 2010. Investigations into the quality of life experienced by these survivors have therefore become necessary if these survivors are to be effectively managed through their course of cancer.

The increase in the number of cancer survivors has opened up a relatively new avenue of cancer research termed Cancer Survivorship Research. Cancer Survivorship Research seeks to investigate the physical, functional and psychosocial consequences of cancer. Despite advances made in survivorship research, gaps remain in our knowledge concerning the ability of the cancer survivor to reintegrate into life and function at pre-cancer levels. These knowledge-gaps are especially true for head and neck cancer patients as demonstrated by the paucity of studies in the literature evaluating the functional and psychosocial consequences of cancer in this cohort. This is a significant short-coming especially since head and neck cancer patients are at increased risks for adverse consequences due to their advanced age at the time of cancer diagnosis, comorbidity burdens and substantial history of alcohol or tobacco use.

This study will evaluate the functional and cognitive changes that occur in head and neck cancer patients as a result of cancer treatment, in an attempt to understand the consequences of cancer treatment on the quality of life experienced by these survivors.

Our study will use self-report questionnaires, neurocognitive assessments and novel performance-based assessments to evaluate functional and cognitive health status at two time-points:

1. At Baseline (before any cancer treatment modality)
2. After the first stage of cancer therapy (chemotherapy, radiation or surgery)

Assessments to be utilized include the Center for Epidemiologic Studies Depression Scale (CES-D), University of Alabama Life Space Assessment Aids form (LSA Aids), Dysexecutive Questionnaire (DEX), Katz Index of Activities of Daily Living (ADLs), Lawton Index of Instrumental Activities of Daily Living (IADLs), University of Alabama Life Space Assessment (LSA), Short Blessed Test (SBT), Short Physical Performance Battery (SPPB), Adult Comorbidity Evaluation-27 (ACE-27), and the Delis Kaplan Executive Function Scale (DKEFS) - Sorting task, Color Word Interference task, and Trail Making task.

Participants will also be assessed using the Executive Function Performance Test (EFPT). The EFPT is a performance-based measure of cognitive function developed at the Program for Occupational Therapy at Washington University School of Medicine that assesses (under direct observation) the amount of assistance needed by participants to complete five basic tasks essential for self-maintenance and independent living. The tasks include hand-washing, cooking, using the telephone, taking medications and paying bills.

Head and Neck cancer patients will undergo these comprehensive assessments at each of the two time-points, allowing for the ability to follow changes in function and cognition over the course of cancer therapy. Statistical analyses will be performed with the SAS® software version 9.1.3 to obtain descriptive statistics and to investigate statistically-significant changes in functional and cognitive health status between the time-points evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 40 years of age or older.
* Subjects must be able to read, write and speak English fluently.
* Subjects must be newly diagnosed with head and neck squamous cell cancer.
* Subjects must not have already had treatment for this cancer diagnosis.
* Subjects must be anticipated to receive at least one of the following types of therapy: surgery, chemotherapy or radiation.

Exclusion Criteria:

* Subjects with prior cancer diagnoses who have evidence of active disease.
* Subjects who have received cancer treatment within the past year.
* Subjects who have received chemotherapy or radiation treatment within the past year (for any disease state).
* Life expectancy of less than 3 months.
* Subjects with melanoma or other non-squamous cell cancer.
* Subjects who score >9 on Short Blessed Test (SBT) at baseline.
* Subjects who are unable to complete all of the required forms and tasks at baseline, either because of cognitive deficits or physical limitations.
* Any medical condition the PI determines to affect safe study participation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the Washington University Physicians Faculty Practice clinics of Adult Otolaryngology, Medical Oncology and Radiation Oncology
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Functional and Cognitive health status | At the time of cancer diagnosis and Within 1 month of cancer therapy

SECONDARY OUTCOMES:
Assess the effectiveness of novel performance-based tests in detecting subtle functional and cognitive health status changes | At the time of cancer diagnosis and Within 1 month of cancer therapy

CONTACTS AND LOCATIONS:
Overall Officials: Oluwafunmilola T Okuyemi, MD, Principal Investigator — Washington University School of Medicine; Jay F Piccirillo, MD, FACS, Study Director — Washington University School of Medicine
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Washington University School of Medicine, St Louis, Missouri